CLINICAL TRIAL: NCT07245576
Title: A Study to Evaluate the Accuracy of Primary Care Diagnosis Using Oscillometry and Fractional Exhaled Nitric Oxide for Asthma and COPD Versus Specialist Diagnosis in Patients With Suspected Asthma or COPD
Brief Title: Assess Accuracy of Primary Care Asthma and COPD Diagnosis Using Oscillometry and FeNO vs Specialist Diagnosis
Acronym: Care4All
Status: Not yet recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D2287R00214
Record Dates: First submitted 2025-10-06; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Asthma; COPD
Keywords: Asthma; COPD; Oscillometry; spirometry; Fractional Exhaled Nitric Oxide Test - FeNO; Chronic Obstructive Pulmonary Disease - COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Current diagnostic methods for asthma and chronic obstructive pulmonary disease mostly depend on pulmonary function tests, especially spirometry. While spirometry is a foundational tool, its diagnostic accuracy is often limited by the patient's ability to perform forceful breathing maneuvers, as well as technical and reproducibility challenges, and the need for proper equipment and training. These constraints can compromise effective diagnosis of asthma and COPD in primary care settings. Prompt and accurate diagnosis by primary care physicians is essential for better patient outcomes. Although variable airflow limitation often measured as a change in FEV1 after bronchodilator is a hallmark of asthma, inconsistencies in test quality and reversibility criteria create challenges in distinguishing asthma from COPD. These complexities highlight the need for alternative diagnostic tools beyond traditional spirometry.

This observational study is designed to evaluate the diagnostic accuracy and technical feasibility of using oscillometry and FeNO testing in primary care for suspected asthma and COPD, compared to conventional specialist-based diagnostics. The study will be conducted across 6 countries in the MEA, Asia, and Latin America, with two hospital sites per country. Primary care physicians will be trained in oscillometry and FeNO testing using standardized protocols and tools such as the Ambulatory Lung Diagnosis System following GINA and GOLD guidelines. Eligible patients will provide consent, complete a history and symptom questionnaire, and undergo primary care-based assessment for a provisional diagnosis. If specialist assessment cannot occur the same day, it will be done within three days. No follow-up visits are planned. Study outcomes will inform the feasibility and accuracy of integrating these methods into routine care, aiming to improve the early and reliable diagnosis of asthma and COPD.

DETAILED DESCRIPTION:
Diagnosis of asthma and chronic obstructive pulmonary disease (COPD) currently relies heavily on pulmonary function tests (PFTs), with spirometry as the core method. However, the effectiveness of spirometry is closely linked to patients' ability to perform maximal, forceful breathing maneuvers. This poses difficulties for individuals with varying physical capacities, leading to challenges in test use, result interpretation, and reproducibility. Such limitations often require skilled specialists, which may not be available in all settings, especially in primary care.

Primary care providers are the initial interface for patients with respiratory symptoms, tasked with rapidly evaluating and diagnosing conditions during brief patient interactions. Early diagnosis of asthma and COPD is crucial, yet spirometry standards-such as those set by the European Respiratory Society and American Thoracic Society-often cannot be met in primary care due to resource and expertise constraints. Operational barriers, including equipment costs, maintenance, staff training, and integration into routine practice, further hinder widespread adoption of spirometry.

Adding to the complexity, variable bronchodilator responsiveness complicates the differential diagnosis of obstructive airway diseases. Traditional reversibility criteria based on FEV1 changes following bronchodilator administration may be unreliable, reducing their diagnostic utility for distinguishing asthma from COPD and highlighting the need for multidimensional approaches.

Oscillometry is emerging as a promising alternative or adjunct to spirometry. It is a non-invasive method capable of detecting airway resistance and reactance, which can reveal early functional changes in asthma and COPD-even before clinical symptoms appear. Oscillometry is valuable for monitoring disease progression, assessing bronchodilator response, and may be more sensitive for small airway dysfunction, especially in patients with normal or slightly impaired lung function.

Measurement of fractional exhaled nitric oxide (FeNO) is another innovative technique. As a marker for T-helper 2 cell-mediated airway inflammation, FeNO can enhance the diagnosis and monitoring of asthma. Guidelines recommend FeNO thresholds for diagnosis and management, adding an objective layer to clinical decision-making. International guidelines advise integrating FeNO and additional objective tests, such as eosinophil counts, with standard PFTs to support asthma diagnosis.

Addressing the considerable unmet need for earlier identification of asthma and COPD, a multicenter, multinational, cross-sectional study has been designed to evaluate the technical feasibility and diagnostic accuracy of oscillometry and FeNO testing in primary care. Conducted across six countries in the Middle East and Africa, Asia, and Latin America, the study will systematically compare primary care-based diagnosis using combined oscillometry and FeNO testing with conventional specialist-led diagnostics.

Patients with suspected asthma or COPD will be enrolled from outpatient departments during a six-month recruitment period. Participating primary care physicians will be trained according to Global Initiative for Asthma (GINA) and Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines, and equipped with tools such as the Ambulatory Lung Diagnosis System. Recruitment will avoid sites biased toward severe cases, ensuring a representative patient population. Provisional diagnoses will be established via history, symptom questionnaires, and results of oscillometry and FeNO testing; where immediate specialist assessment is not feasible, patients will return within three days for further evaluation. No follow-up visits are planned. The study aims to inform clinical practice by clarifying the feasibility and effectiveness of integrating these innovative diagnostic methods into primary care, with the goal of facilitating earlier and more reliable identification of asthma and COPD.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the study if all the following criteria apply and after providing written informed consent:

Suspected asthma (asthma group)

1. Patients ≥ 18 years old or with legal age of consent in the jurisdiction in which the study is taking place, at the time of signing the ICF.
2. Patients presenting with symptoms of wheezing, cough, chest tightness, shortness of breath, but without a clinically confirmed diagnosis of asthma.

Suspected COPD (COPD group)

1. Patients ≥ 40 years old at the time of signing the ICF.
2. Patients presenting with symptoms of dyspnea, chronic cough or sputum production, but without a clinically confirmed diagnosis of COPD.

Exclusion Criteria:

Patients are excluded from the study if any of the following criteria apply:

1. Prior diagnosis of COPD or asthma.
2. Use of ICS in the last 6 months or use of oral corticosteroids in the last 3 months.
3. Any diseases that influence lung function result such as lung cancer, pneumonia, active pulmonary tuberculosis, pulmonary embolism, and interstitial lung disease.
4. Any history of recent surgery that affects lung function results, including but not limited to thoracotomy surgery, pneumothorax surgery, and thoracic drainage.
5. Contraindication to spirometry or oscillometry test, or allergy to bronchodilator.
6. Currently pregnant or breast-feeding women.
7. If the investigator judges that the patient is unlikely to comply with study procedures, restrictions, and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total of 600 patients (approximately 300 suspected asthma patients and 300 suspected COPD patients) will be enrolled in this study. The patients will be enrolled in asthma or COPD groups in 1:1 ratio at site-level. Each site will enroll 50 patients (approximately 25 suspected asthma and 25 suspected COPD).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-11-14 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of primary care asthma/COPD diagnosis using oscillometry (ALDS: R5, R20, R5-R20, X5, Ax) plus FeNO ≥50 ppb (Fenom PRO®/ALDS Pro) vs specialist gold standard; metrics: Cohen's kappa, agreement, sensitivity, specificity in overall, asthma, COPD | 1 to 3 days
  Primary care diagnosis uses a diagnostic algorithm combining oscillometry and FeNO. Oscillometry: Ambulatory Lung Diagnosis System (ALDS) parameters-respiratory system resistance at 5 Hz (R5), resistance at 20 Hz (R20), difference R5-R20, reactance at 5 Hz (X5), and area of reactance (Ax). FeNO: measured with Fenom PRO® or ALDS Pro devices, using a diagnostic cut-off of ≥50 ppb.
  Specialist care diagnosis is the comparator: Gold Standard Specialist Care Diagnosis established through standard clinical practice, including pulmonary function tests, spirometry, physiological tests, imaging, laboratory tests, and bronchial provocation tests.
  Accuracy will be quantified using Cohen's Kappa coefficient, Percentage Agreement, Sensitivity, and Specificity. The analysis will be conducted in the overall population, the asthma group, and the COPD group.

SECONDARY OUTCOMES:
accuracy and agreement between asthma or COPD diagnoses made in primary care with provisional diagnoses derived exclusively from patient history compared to specialist settings diagnosis | 1 to 3 days
  To evaluate the accuracy and agreement between asthma or COPD diagnoses made in primary care with provisional diagnoses derived exclusively from patient history compared to specialist settings diagnosis

OTHER OUTCOMES:
Healthcare provider satisfaction with primary care diagnostic tests (oscillometry and FeNO) as measured by a 5-point Likert scale (ranging from 1 'not satisfied at all' to 5 'very satisfied', where higher scores indicate greater satisfaction) | 1 to 3 days
  This directly measures the satisfaction scores or experience rating (as per Protocol Section 2, Table 1 and Section 3.1.1.1) using the specified 5-point Likert scale, including its range and interpretation, addressing both Major and Advisory Issues
Primary care provider confidence in their diagnosis (for this patient) as measured by a 5-point Likert scale (ranging from 1 'not at all confident' to 5 'extremely confident', where higher scores indicate greater confidence) | 1 to 3 days
  This measures the confidence scores (as per Protocol Section 2, Table 1 and Section 3.1.1.1) of primary care providers in their diagnostic assessment using the specified 5-point Likert scale, including its range and interpretation.
Specialist care provider experience with the diagnostic process at secondary care as measured by a 5-point Likert scale (ranging from 1 'very challenging' to 5 'very straightforward', where higher scores indicate a more straightforward experience) | 1 to 3 days
  This measures the experience scores (as per Protocol Section 2, Table 1 and Section 3.1.1.1) of specialist care providers with the diagnostic process, utilizing the specified 5-point Likert scale, including its range and interpretation.

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home